CLINICAL TRIAL: NCT04237597
Title: Pharmacokinetic Drug-Drug Interaction Study Between K-877 and CSG452 in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kowa Research Institute, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K-001-001
Record Dates: First submitted 2020-01-16; First posted 2020-01-23 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Healthy
MeSH Terms: interventions — K-877 compound; 6-((4-ethylphenyl)methyl)-3',4',5',6'-tetrahydro-6'-(hydroxymethyl)spiro(isobenzofuran-1(3H),2'-(2H)pyran)-3',4',5'-triol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- K-877 & CSG452 (Experimental): K-877 Single dose on Day 1 and Day 15 CSG452 Repeat dose on Day 2 Through Day 15
  Interventions: Drug: K-877; Drug: CSG452

INTERVENTIONS:
Drug: K-877 — K-877 tablets
Drug: CSG452 — CSG452 tablets

SUMMARY:
A study to compare the pharmacokinetic(s) of K-877 and CSG452 when each drug is administered alone and when both are administered together.

ELIGIBILITY:
Inclusion Criteria:

* Subject provides written informed consent before any study-specific evaluation is performed.
* Subject is a healthy adult male or female volunteer between the ages of 18 and 45 years, inclusive, at Screening.
* Subject has a BMI of 18 to 30 kg/m2, inclusive, at Screening.
* Subject meets all other inclusion criteria outlined in the clinical study protocol

Exclusion Criteria:

* Subject has clinically relevant abnormalities at Screening or at Check-in assessments.
* Subject is pregnant or breastfeeding or intends to become pregnant within 30 days after the last dose of study drug.
* Subject does not meet any other exclusion criteria outlined in the clinical study protocol.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-12-17 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-03-04 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) | 0 to 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- PPD Development. LP, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided